CLINICAL TRIAL: NCT01328106
Title: A Single-Arm, Open-Label, Multi-Center Study to Investigate the Objective Response Rate, Safety, and Pharmacokinetics of GSK1120212, a MEK Inhibitor, in Subjects With Metastatic Uveal Melanoma or With Mutation-Positive GNAQ or GNA11 Metastatic Melanoma
Brief Title: Efficacy and Safety Study of GSK1120212, a MEK Inhibitor, in Subjects With Uveal Melanoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was cancelled by the sponsor prior to initiation of study enrollment. No subjects were accrued.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 114091
Record Dates: First submitted 2010-03-18; First posted 2011-04-04 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: GNA11 Mutation-positive Metastatic Melanoma; GNAQ Mutation-positive Metastatic Melanoma; Cancer; Metastatic Uveal Melanoma
MeSH Terms: conditions — Neoplasms; Uveal Melanoma | interventions — trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: GSK1120212

INTERVENTIONS:
Drug: GSK1120212 — Repeating oral dose

SUMMARY:
The purpose of this study is to determine whether GSK1120212, a MEK inhibitor, is an effective and safe treatment for cancer subjects with metastatic uveal melanoma and mutation-positive GNAQ or GNA11 metastatic melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of metastatic uveal melanoma or previously documented mutation-positive GNAQ or GNA11 metastatic melanoma not previously treated with a MEK inhibitor.
* Provide archival tumor tissue or, if tissue blocks are not available, undergo fresh tumor biopsy prior to enrollment.
* The patient has a radiographically measurable tumor.
* ECOG performance status 0, 1, or 2.
* The patient is able to swallow and retain oral medication.
* Life expectancy of at least 4 months.
* Toxicities from previous anti-cancer therapy (except alopecia) are recovered (Grade 1 or less) at the time of enrollment.
* The patient has adequate organ and bone marrow function.
* Sexually active patients must use medically acceptable methods of contraception during the course of the study.
* Female patients of childbearing potential must have a negative serum pregnancy test at screening.

Exclusion Criteria:

* The patient has had any of the following within 21 days of starting study drug or anticipates the need for any of the following during the course of study treatment: chemotherapy, immunotherapy, biologic therapy, hormone therapy, major surgery, or tumor embolization.
* The patient has received experimental therapy within 21 days of starting study drug.
* The patient has received nitrosourea or mitomycin C within 42 days of starting study drug.
* The patient has received any herbal medications or palliative radiotherapy within 14 days of starting study drug.
* The patient is currently receiving anticoagulation therapy that is not well controlled.
* Ongoing or newly diagnosed eye abnormality other than symptoms due to uveal melanoma.
* History of retinal vein occlusion or central serous retinopathy.
* Current severe, uncontrolled systemic disease.
* History of leptomeningeal disease or spinal cord compression secondary to metastasis.
* Brain metastasis, unless previously treated with surgery, whole-brain radiation or stereotactic radiosurgery and the disease has been stable for at least 3 months without steroid use or on a stable dose of steroids for at least 1 month prior to starting study drug. Stability of brain metastases must be confirmed with imaging.
* The patient has a concurrent, active hematological malignancy or other solid tumor malignancy.
* History of clinically significant cardiac or pulmonary dysfunction.
* Allergy or hypersensitivity to components of the GSK1120212 formulation.
* The patient is pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-11; Primary Completion 2011-08 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Objective response rate as assessed by RECIST v1.1 | At least 12 weeks after initiating study treatment

SECONDARY OUTCOMES:
Duration of response, progression free survival, overall survival | Through study completion or early study discontinuation
Safety, tolerability, and population pharmacokinetic parameters | Through study completion or early study discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline